CLINICAL TRIAL: NCT01503697
Title: The Role of the Novel 99mTc-NC100692 Tracer in Patients at High Risk or Known Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, director, R&D Division, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-11-EE-262-CTIL
Record Dates: First submitted 2012-01-01; First posted 2012-01-04 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer; Tumor Angiogenesis
Keywords: Breast Cancer; High Risk; Imaging; Angiogenesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Technetium-99m NC100692 Injection is under development as a diagnostic radiopharmaceutical for targeting angiogenesis associated with diseases such as primary and metastatic cancer, and for targeting active fibrosis in cardiac diseases such as developing heart failure and developing hypertrophic cardiomyopathy.

A principle goal of imaging is identification of disease processes early in their development, at times prior to symptoms. In cancer, angiogenesis is essential for a tumour to exceed approximately 1-2 mm3 in size.As markers of angiogenesis are often expressed early in the growth of a tumour it is postulated that imaging of angiogenesis can assist in early diagnosis of cancer, relapse or spread, and monitoring response to therapy.

Technetium-99m NC100692 Injection will be tested on 3 populations of pts:

1.30 patients at high risk For breast cancer 2.30 patients with breast cancer 3.15 patients with locally advanced breast cancer undergoing treatment.

DETAILED DESCRIPTION:
Angiogenesis is the formation of new blood vessels from the existing vascular bed. Certain integrins are upregulated while angiogenesis and myocardial fibrogenesis. Therefore, targeting an integrin with an imaging agent can be potentially useful for the early diagnosis of angiogenesis and/or fibrogenesis of malignant processes and myocardial remodelling.

Trail design

Arm 1:

Study cohort will include 30 patients. After the IV injection of 630-700 MBq 99mTc-NC100692 each breast will be imaged in CC and oblique views using the MBI system. Scintigarphic findings will be correlated with tissue diagnosis and or/ imaging and clinical follow- up of at least 6 months as well as with MRI, if performed, in order to determine the PPV and the NPV of the technology of MBI with labeled NC100692 for detection of tumors and differentiating benign and malignant breast lesions.

Arm 2 :

Study cohort will include 30 patients with breast cancer referred for 18-FDG PET-CT for staging or re-staging. In addition to the PET-CT study, scintimammography using the MBI system and whole-body scintigraphy using the Infinia gamma-camera will be performed after the IV injection of 630-700 MBq 99mTc-NC100692. Imaging with 99mTc-NC100692 will be take place first followed by 18-FDG PET-CT, on the same day.

Detection of the primary tumor, lymph nodes and remote metastasis by the various modalities and tracers will be correlated.

Arm 3:

Study cohort will include 15 patients with locally advanced breast cancer. Patients will undergo scintimammography with the MBI system (for the breast) and SPECT of the axilla and thorax (for regional lymph nodes) with the Infinia gamma camera, after the IV injection of 630-700 MBq 99mTc-NC100692 prior to treatment and at its end. The results of the follow-up studies will be correlated with histological findings in patients referred for surgery and with MRI in others.

Prior to the exam, patients will answer a detailed questionnaire about medical and family history,findings on other imaging modalities and,therpy.

The patient will be guided by the study coordinator before answering the questionnaire Reading of the 99mTc-NC100692 studies will be in a blinded mode to other imaging data, separately by two nuclear medicine experts and then in consensus. Mammography, US and MRI will be reviewed by a breast imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients with unknown breast cancer but unclear lesions in the breast on other modalities or patients at high risk for breast cancer (BRCA, familial)- Arm 1
* patients with breast cancer referred for 18-FDG PET-CT for staging or re-staging- Arm 2
* Study cohort will include 15 patients with locally advanced breast cancer. Patients will undergo imaging prior to treatment and at its end- Arm 3
* Written signed informed consent to participate in the study.
* Patients not pregnant or lactating.

Exclusion Criteria:

* Patients with breast cancer who do not fall into one of the three study arms.
* Pregnant or lactating females.
* Participation in another investigational study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigating the diagnostic accuracy of NC100692kit in three patient populations:
  Arm 1.Patients with unknown breast cancer but unclear lesions in the breast or other modalities or patients at high risk for breast cancer (BRCA, familial) Arm 2. Staging and re-staging in patients with breast cancer. Arm 3. Monitoring response to neo-adjuvant chemotherapy in patients with locally advanced breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2012-01

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Einat Even-Sapir Weizer, MD, PhD, Principal Investigator — Head, Department of Nuclear Medicine,Tel Aviv Sourasky Medical Center
Locations (1):
- Department of Nuclear Medicine,Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Buerkle MA, Pahernik SA, Sutter A, Jonczyk A, Messmer K, Dellian M. Inhibition of the alpha-nu integrins with a cyclic RGD peptide impairs angiogenesis, growth and metastasis of solid tumours in vivo. Br J Cancer. 2002 Mar 4;86(5):788-95. doi: 10.1038/sj.bjc.6600141. PMID 11875744
- [Background] Folkman J. What is the evidence that tumors are angiogenesis dependent? J Natl Cancer Inst. 1990 Jan 3;82(1):4-6. doi: 10.1093/jnci/82.1.4. No abstract available. PMID 1688381